CLINICAL TRIAL: NCT03469440
Title: Goal Directed Therapy Aiming to Optimise Oxygen Central Venous Saturation in Children Undergoing Cardiac Surgery: a Randomized and Prospective Clinical Trial
Brief Title: Goal Directed Therapy Aiming to Optimise Oxygen Central Venous Saturation in Children Undergoing Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Associate Professor of Anesthesiology Departament, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3988.13.113
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; C.Surgical Procedure; Cardiac
Keywords: lactate; central venous saturation; Pediatric Cardiac Surgery
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed therapy (Active Comparator): Patients randomized to this group will be monitoring by continuous central venous oxygen saturation. Central venous oxygen saturation will be targeted higher than 65% in non-cyanogenic patients and 55% in cyanogenic.
  Interventions: Other: Continuous central venous oxygenation monitoring
- Standard protocol (Other): The control group will keep the standard therapy.
  Interventions: Other: Standard protocol

INTERVENTIONS:
Other: Continuous central venous oxygenation monitoring — Central venous oxygen saturation will be targeted higher than 65% in non-cyanogenic patients and 55% in cyanogenic.
  * First, isotonic crystalloid, 10 up to 20 mL/kg, will be administered in boluses to achieve continuous central venous oxygen saturation higher than 65% in non-cyanogenic and 55% in cyanogenic.
  * Second, if not achieved with fluid administration, will be targeted by initiating and titrating inotropics (dobutamine or milrinone). If the mean arterial pressure is lower than 50 mm Hg will be associated epinephrine.
  * If the ScvO2 is lower than 65% in non-cyanogenic and 55% in cyanogenic and the hemoglobin was lower than 8g/dl, red blood cells (20mL/Kg) will be transfused to achieve a hemoglobin level of at least 8g/dL.
  Arms: Goal-directed therapy
Other: Standard protocol — The control group will keep the standard therapy to achieve mean arterial pressure higher than 50mmHg, central venous pressure 8 to 12 mmHg, urinay debit higher than 0,5ml/kg/h, hemoglobin higher or equal than 8g/dL, arterial oxygen saturation higher or equal than 92% in non-cyanogenic and 80% cyanogenic, central venous oxygen saturation higher or equal than 65% in non-cyanogenic and 55% in cyanogenic.
  Arms: Standard protocol

SUMMARY:
The purpose of this study is evaluate goal-directed therapy with continuous central venous saturation compared to standard therapy in children undergoing cardiac surgery.

DETAILED DESCRIPTION:
Pediatric patients undergoing cardiac surgery are at risk for adverse clinical outcomes due a inadequate tissue perfusion. Recent studies have been demonstraded which the monitorization of continuos central venous saturation could be benneficial. There is evidence that monitoring continues venous oxygen saturation (ScvO2) can be beneficial in patient outcomes, guided by ScvO2 therapy has been associated with improved outcomes in resuscitation of critically ill patients with sepsis and after congenital heart surgery complexa. The early detection and treatment of tissue hypoxia can prevent morbidity and mortality. tissue hypoxia may be a result of the imbalance between supply (DO2) and oxygen consumption (VO2). If the fault supply, oxygen consumption is maintained by increased oxygen extraction resulting in decreased central venous oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery with cardiopulmonary bypass
* Written informed consent

Exclusion Criteria:

* Cardiac arrhythmia
* Emergency operation
* Hemodynamic instabillty (norepinephrine higher than 1 mcg/kg/min)
* Neoplasia
* Heart transplant
* Participation in another study

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lactate clearance | at the beginning of surgery up to 24 hours after surgery
  ([lactate initial - lactate delayed]/lactate initial) ×100%

SECONDARY OUTCOMES:
Length of Mechanical ventilation | within 30 days after cardiac surgery
  hours
Vasopressors and inotropic therapy | within 30 days after cardiac surgery
  hours
Cardiac complications | within 30 days after cardiac surgery
  Low cardiac output syndrome , vasoplegia
Renal complications | within 30 days after cardiac surgery
  Assess by pediatric RIFLE
Infection | within 30 days after cardiac surgery
  Pneumonia, bloodstream, urinary, surgical site and/or sepsis
Length of ICU stay | within 30 days after cardiac surgery
  days
Length of hospital stay | within 30 days after cardiac surgery
  days

CONTACTS AND LOCATIONS:
Overall Officials: Flavio M Ferreira, Phd, Principal Investigator — HCFUSP
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No